CLINICAL TRIAL: NCT01194362
Title: A Study to Establish Genomic Bio Signatures of Ascending Aortic Aneurysms in Patients With Bicuspid and Tricuspid Aortic Valve Disease With Aortic Stenosis
Brief Title: A Study to Identify Differences in Gene Expression in Patients With Bicuspid and Tricuspid Valve Disease
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 010-161
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Aortic Valve Disease
Keywords: aortic valve disease; gene expression
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 45 specimens collected from BAV patients
- 45 specimens collected from TAV patients
- 15 specimens collected from CABG pts

SUMMARY:
For this study, blood and tissue samples will be collected in order to perform genetic testing to help researchers gather information about this disease and how and why it affects some patients more than others.

DETAILED DESCRIPTION:
The cause of bicuspid aortic valve (BAV) and its associated co morbidities is unknown. There is, however, evidence supporting a genetic cause for the BAV, Pedigree analysis of familial clustering initially directed investigators to a genetic cause of BAV. Subsequent studies on BAV patients using linkage analysis have demonstrated high heritability.

Early identification of those patients with BAV disease who are at risk for ascending aneurysm formation and its complications may allow early intervention to prevent rupture, dissection and emergent cardiac surgery in at risk patients. Conversely, identification of those patients with BAVs not at risk for aortic aneurysm formation would delineate which patients do not need close follow up of aortic size or prophylactic ascending aortic replacement at time of aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = to 18 years of age
* Presenting with aortic stenosis and to undergo elective aortic valve replacement or repair with or without aortic aneurysm dilation repair
* Able to sign informed consent document

Exclusion Criteria:

* Patients unable to provide informed consent for any reason
* Patients with predominant aortic regurgitation valve disease
* Patients with other known connective tissue disorders (such as Marfan's Syndrome, Ehlers-Danlos Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital facility
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2010-06-20 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Determine differences in genetic expression profiles using mRNA transcriptional analysis | 12 month
  Determine differences in genetic expression profiles using mRNA transcriptional analysis in the three groups: subjects with bicuspid aortic valves with aortic stenosis, subjects with tricuspid aortic valves with stenosis, and subjects without aortic valve disease.

SECONDARY OUTCOMES:
Determine differences in the association between genetic expression profiles and aortic dilation in the two aortic valve disease groups. | 12 months
  Determine differences in the association between genetic expression profiles and aortic dilation (in cm) among: subjects with bicuspid aortic valves and subjects with tricuspid aortic valves with aortic stenosis.
Determine the association between expression of inflammatory markers/impaired response to oxidative stress and stenotic aortic valve disease. | 12 months
  Determine differences between expression of inflammatory markers/impaired response to oxidative stress and stenotic aortic valve disease among: subjects with bicuspid aortic valves and subjects with tricuspid aortic valves with aortic stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: William Brinkman, MD, Principal Investigator — The Heart Hospital Baylor Plano
Locations (1):
- The Heart Hospital Baylor Plano, Plano, Texas, United States